CLINICAL TRIAL: NCT01808976
Title: Can Mental Health Apps Work in the Real World? A Feasibility Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joaquin Anguera, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34MH100466 (NIH)
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: MDD
MeSH Terms: interventions — Biological Evolution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Evolution (Active Comparator): This app is designed to be a cognitive training game that conditions the CCN. This is done by having participants play a multitasking game that targets their perceptual discrimination abilities, selective attention, and visuomotor tracking skills. At the first session, participants will be directed to an initial assessment of each of these cognitive control skills in a single task and dual-task setting (a total of 3 different diagnostics, described below). Each week, this diagnostic phase will reflect the training paradigm they will encounter for that week, as each week the perceptual and tracking challenges will increase.
  Interventions: Behavioral: Evolution
- Problem Solving Therapy (Experimental): This app is based on the social problem solving protocol developed by Nezu and D'Zurilla . The app begins with explaining the PST steps. Participants are informed that they can learn each step one session at a time, or they can chose to learn all the steps at once. After each step completed, participants are asked if they want to continue onto the next step or save it for the next session, thus the app tailors itself to the users ability to absorb new information.
  Interventions: Other: Problem Solving Therapy
- Basic health push app (Active Comparator): This app provides daily suggestions for overcoming depressed mood and allows users to track their mood, using the 0-9 scale available for all three apps. In the first app session, participants are given a general education about depression and its known causes and consequences. Participants are told that to overcome mood problems, they must engage in one mood improvement strategy a day and that the app will suggest one to try each day.
  Interventions: Behavioral: Basic health push app

INTERVENTIONS:
Other: Problem Solving Therapy — this is a mobile app that participants use to solve problems. It will guide participants through a stepwise process for identifying a means for creating action plans.
  Arms: Problem Solving Therapy
Behavioral: Evolution — This is a therapeutic video game that targets the cognitive control network, associated with depression. Participants are expected to play the game daily for 20 minutes over 4 weeks.
  Arms: Evolution
Behavioral: Basic health push app — This is an app that send daily tips for improving your mood.
  Arms: Basic health push app

SUMMARY:
Over two million people in the US download health apps onto their smartphones and tablets, with the intent of improving their quality of life. Despite widespread use of these apps, there is relatively little information regarding app user access (do users download health apps and use them more than once), app user engagement (do users follow the app protocols) and app impact on mood, cognition and daily functioning. Our long-term goal is to conduct a future randomized controlled trial investigating access, engagement and impact of two types of mental health apps, apps based on evidence-based therapeutic principles (i.e.: Problem Solving Therapy) and apps based on cognitive neuroscience principles of depression (i.e.: a cognitive training game called Evolution) and compare both to an information only app. Our intent is to conduct this study entirely on mobile devices, in order to investigate access, engagement, and impact in an ecologically valid manner. The purpose of this pilot study is to test the feasibility of conducting our future randomized controlled trial comparing three mobile mental health apps for the management of depressed mood, improvement of cognitive control, and improvement in activities of daily living in people aged 18 and older. Recruitment, consent, randomization, app use and outcome assessment will be conducted entirely on mobile devices. We will recruit 150 people through four different recruitment avenues to determine which avenue results in the most representative sample of our target population (people 18 and older who have symptoms of depression that are interfering with their quality of life). We will also determine the number we need to recruit to have a final sample of 150 people willing to be randomized between the 3 apps and complete an 12-week study of app impact on mood, cognition and function. This pilot will provide information on the completeness of data from a study conducted in this manner, and uncover any other challenges we may face by using mobile devices for data collection, and if we will find differential drop out between app type (e.g.: will more people stop using of the information only app prematurely?). Although we will not have sufficient statistical power to answer questions about comparative effectiveness between the apps, we plan to explore relationships between sample demographics, app use, and improvement in cognitive control on improvements in mood and function.

DETAILED DESCRIPTION:
Participants will be recruited nationally from a variety of on-line sources. Participants will complete a breif on-line survey and then randomized to one of three mobile apps for depression. Participants are expected to use the apps for 4 weeks, complete daily ratings of mood, as well as complete 4 comprehensive assessments on their smart devices at weeks 1, 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* must own smart device (iPhone or ANDROID + iPAD)
* a total score of 5 or greater on the PHQ-9; OR a score of 2 or greater on at least one of the first two PHQ-9 items AND a score of 2 or greater on the 10th PHQ-9 item
* English speaking* (* as of 12/2016: this arm is closed)
* Spanish speaking (1st or second language)

Exclusion Criteria:

* below 18 years or older
* does not own a smart device
* a total score of less than 5 on the PHQ-9
* less than a score of 2 on the first two PHQ-9 items and less than 2 on the 10th PHQ-9 item

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Sheehan Disability Assessment Scale | Up to 3 weeks
  Assesses functional impairment in three inter-related domains; work/school, social and family life.
Patient Global Improvement Scale | Up to 3 weeks
  A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Patient Health Questionnaire | Up to 3 weeks
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment.
Sheehan Disability Assessment Scale | Week 8
  Assesses functional impairment in three inter-related domains; work/school, social and family life.
Patient Global Improvement Scale | Week 8
  A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Patient Health Questionnaire | Week 8
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment.
Sheehan Disability Assessment Scale | Week 12
  Assesses functional impairment in three inter-related domains; work/school, social and family life.
Patient Global Improvement Scale | Week 12
  A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Patient Health Questionnaire | Week 12
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Web-based; log onto www.brightenstudy.com/spa for details, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to release data for sharing once the study is complete.

REFERENCES:
- [Derived] Renn BN, Pratap A, Atkins DC, Mooney SD, Arean PA. Smartphone-Based Passive Assessment of Mobility in Depression: Challenges and Opportunities. Ment Health Phys Act. 2018 Mar;14:136-139. doi: 10.1016/j.mhpa.2018.04.003. Epub 2018 Apr 18. PMID 30123324
- [Derived] Pratap A, Renn BN, Volponi J, Mooney SD, Gazzaley A, Arean PA, Anguera JA. Using Mobile Apps to Assess and Treat Depression in Hispanic and Latino Populations: Fully Remote Randomized Clinical Trial. J Med Internet Res. 2018 Aug 9;20(8):e10130. doi: 10.2196/10130. PMID 30093372